CLINICAL TRIAL: NCT00984230
Title: A New Adaptive Feeding Plan for Newborns: Effects on Gut Maturity and Gut Microbiota
Brief Title: A New Adaptive Feeding Plan for Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 07.22.INF
Record Dates: First submitted 2009-09-10; First posted 2009-09-25 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Infant Nutrition
Keywords: Infant Formula; Gut
MeSH Terms: interventions — Busulfan; Lactoferrin; Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Breastfeeding (Reference) (No Intervention)
- Basic starter formula: BSF (Active Comparator)
  Interventions: Other: BSF
- BSF + Lactoferrin + Probiotics + OS (Experimental)
  Interventions: Other: BSF + Lactoferrin + Probiotics + OS
- BSF + Lactoferrin + Probiotics (Experimental)
  Interventions: Other: BSF + Lactoferrin + Probiotics

INTERVENTIONS:
Other: BSF — feeding amount according to individual baby need
  Arms: Basic starter formula: BSF
Other: BSF + Lactoferrin + Probiotics — feeding amount according to individual baby need
  Arms: BSF + Lactoferrin + Probiotics
Other: BSF + Lactoferrin + Probiotics + OS — feeding amount according to individual baby need
  Arms: BSF + Lactoferrin + Probiotics + OS

SUMMARY:
The purpose of this clinical trial is to identify the infant formula(s) for which the investigators get the closest gut maturation index compared to the one they get with breastfed babies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborn infant
* Full term infant (≥ 37 weeks gestation; < 42 weeks gestation)
* Birth weight from 2500g to 4500g
* For the formula-fed groups: babies whose mothers elected not to breastfeed at all
* For the breastfed group: babies whose mothers elected to exclusively breastfeed for at least 2 months
* Newborn whose parents / caregivers can be expected to comply with the protocol
* Study explained and written information given
* Informed consent signed

Exclusion Criteria:

* Mother who had antibiotics in the 7 days preceding delivery
* Caesarian section
* Multiple birth
* Congenital illness or malformation that may affect normal growth
* Significant pre-natal and/or post-natal disease
* Newborn participating in another clinical trial

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 186 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
gut maturation : Specific proteins in stools | 3rd day, at 1 week, 2 weeks and 1 month of age

SECONDARY OUTCOMES:
Growth and gut microbiota | At 1 month and 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Pr Picaud, Principal Investigator — Service de Réanimation Néonatale et Néonatologie, Hôpital de la Croix Rousse
Locations (6):
- Department of Pediatrics, Vienna, Austria
- France (4):
  - Service de Réanimation Néonatale et Néonatologie, Hôpital de la Croix Rousse, Lyon
  - Maternité Régionale, Service de Néonatologie, Nancy
  - Service de Néonatologie, Nantes
  - Hôpital Charles Nicolle, Département de Pédiatrie, Rouen
- Alexandra Regional General Hospital, Department of Neonatology, Palaió Fáliro, Athens, Greece